CLINICAL TRIAL: NCT07270666
Title: Pragmatic Pilot Study of ctDNA Informed Immune Checkpoint Inhibitor De-escalation in Advanced/Recurrent Mismatch Repair Deficient (MMR-D)/Microsatellite Instability High (MSI-H) Endometrial Cancer Using Standard of Care Treatments
Brief Title: ctDNA Testing to Inform Standard-of-Care Treatment Decisions in People With Endometrial Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25-337
Record Dates: First submitted 2025-11-26; First posted 2025-12-08 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Endometrial Cancer
Keywords: Stage III with residual disease; Stage IV; Recurrent endometrial cancer after adjuvant therapy only; ctDNA Testing; 25-337
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: This is a pragmatic, pilot study of ctDNA informed, immune checkpoint inhibitor (ICI) de-escalation in advanced/recurrent mismatch repair deficient (MMR-D)/microsatellite instability high (MSI-H) endometrial cancer with a feasibility primary endpoint.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ctDNA-negative group (Experimental): Participants in this group will have negative ctDNA test results at 1 year after they start standard treatment. (Negative results indicate that no cancer DNA is detected in their blood.) Participants in this group will decide with their doctor if they want to stop standard maintenance ICI treatment.
  Interventions: Genetic: ctDNA Testing; Other: Blood draw
- ctDNA-positive group (Experimental): Participants in this group will have positive ctDNA test results at 1 year after they start standard treatment. (Positive results indicate that cancer DNA is detected in their blood.) Participants in this group will continue receiving standard treatment with their doctor.
  Interventions: Genetic: ctDNA Testing; Other: Blood draw

INTERVENTIONS:
Genetic: ctDNA Testing — Patients will undergo ctDNA sampling at the 1-year timepoint using the commercially available Natera SignateraTM test.
Other: Blood draw — at the 1-year timepoint

SUMMARY:
The researchers are doing this study to evaluate the use of circulating tumor DNA (ctDNA) testing in making treatment decisions for advanced/recurrent endometrial cancer that has a change (mutation) in the mismatch repair deficient (MMR-D) gene or microsatellite instability high (MSI-H) gene. The researchers will see how doctors and their patients use the results of ctDNA testing after 1 year of standard chemotherapy and immune checkpoint inhibitor (ICI) treatment to decide whether to continue maintenance ICI treatment past 1 year. The researchers will also look at the health outcomes of people in this study (for example, whether they are cancer free at the end of their participation in the study).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have pathologically confirmed endometrial cancer
* Patients with advanced endometrial cancer
* Stage III with residual disease
* Stage IV
* Recurrent endometrial cancer after adjuvant therapy only
* Patients can have primary or planned interval surgery
* MMR-D on immunohistochemistry OR MSI-H using any commercially available test
* Patients with treated brain metastases are eligible if follow up brain imaging after CNS directed therapy shows no evidence of progression.
* Eligible for standard of care chemotherapy with immune checkpoint inhibitor per treating investigator with no clinical contraindications
* For the up to 10 patients who are allowed to enroll after C1D1 of standard of care treatments, they need to be on treatment with no clinical evidence of disease progression.

  * Patients may have received prior radiation therapy for treatment of endometrial cancer. Prior radiation therapy may have included pelvic radiation therapy, extended field pelvic/para aortic radiation therapy, intravaginal brachytherapy, and/or palliative radiation therapy.
  * Patients may have received prior hormonal therapy for treatment of endometrial cancer.
  * Patients may not have received prior therapy with an anti-PD-1, anti-PD-L1 or anti-CTLA-4 therapeutic antibody or other similar agents.

    * Except for the up to 10 patients who are allowed to enroll after C1D1 of standard of care treatments (chemotherapy and/or immune checkpoint inhibitors) per protocol.
* Age ≥ 18
* Not Pregnant and Not Nursing

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Endometrial Cancer
Enrollment: 30 (Estimated)
Dates: Start 2025-11-25 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
will test the feasibility of ct-DNA | 1 year
  informed de-escalation of standard of care ICI maintenance therapy defined as willingness of patients/providers to stop ICI therapy after 1 year in those with negative ctDNA testing.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Liu, MD, MPH, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (All Protocol Activites), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (All Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (All Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk - Commack (All Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (All Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (All Protocol Activities), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org